CLINICAL TRIAL: NCT06438796
Title: Efficacy and Safety of Blinatumomab Maintenanceafter Allogeneic Hematopoietic Stem Cell Transplantation for High-risk Acute B-lymphoblastic Leukemia: a Multicenter, Open-label, Randomized Controlled Study
Brief Title: Blinatumomab Maintenance After Allo-HSCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TROPHY-ALL01
Record Dates: First submitted 2024-05-23; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: High Risk Acute Lymphoblastic Leukemia
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blinatumomab group (Experimental): Blinatumomab group (Blinatumomab): 9 μg/d intravenously over 24 hours until the end of d14 days of dosing. Repeat every 3 months for a total of 4 courses. (Basis for Dose Selection: The recommended dose of blinatumomab for MRD-negative patients is 9ug/d)
  Interventions: Drug: Blinatumomab
- Control group (No Intervention): Maintenance therapy in the control group was based on the routine maintenance therapy in each center (including but not limited to decitabine, sorafenib, prophylactic DLI, except for all types of CD19 mono- and dual-antibodies and CD22-ADC drugs).

INTERVENTIONS:
Drug: Blinatumomab — Maintenance therapy with Blinatumomab initiation: 90 days to 120 days post-transplantation
  Arms: Blinatumomab group

SUMMARY:
To evaluate the safety and efficacy of Blinatumomab maintenance after allogeneic hematopoietic stem cell transplantation for high-risk acute B-lymphoblastic leukemia.

DETAILED DESCRIPTION:
Blinatumomab is a novel immunological antibody based on BiTE. CD19 is a surface antigen expressed throughout the development of B lymphocytes, making it an ideal target for immunotherapy. Blinatumomab was approved by the FDA for the treatment of adults with relapsed/refractory cancers. Open-label, single-arm, multicenter phase II clinical study (BLAST study) , enrolling 116 adult patients with precursor B-ALL in complete hematologic remission after at least 3 doses of intense chemotherapy but persistently positive for Measurable Residual Disease (MRD) (MRD ≥10-3 ), which is the first ALL international multicenter clinical trial. In August 2022, China's National Medicines and Pharmaceutical Administration (NMPA) Approved Blinatumomab for the treatment of relapsed/refractory precursor B-cell ALL in adults.

Blinatumomab is mostly used for preemptive therapy after post-transplant MRD conversion, and fewer prospective studies have been conducted in the area of maintenance therapy. A prospective single-arm clinical study (NCT02807883) with Blinatumomab as maintenance therapy (up to 4 cycles) after allogeneic transplantation, concluded by MD Anderson in August 2021, had the primary endpoints of safety (acute graft-versus-host disease [aGVHD] and non-relapse mortality [NRM]) and the secondary endpoints of efficacy (PFS, OS, etc.), a total of 23 patients were enrolled in patients who received at least 1 cycle of Blinatumomab, the interval between transplantation and the first cycle of Blinatumomab use was 78 days (44-105), 57% of the patients completed 4 cycles of treatment, the median follow-up was 14.3 months, the 1-year NRM was 0%, the incidence of grade 3-4 aGVHD was 5%, the 1-year OS was 85%, and the 1-year PFS was 71%. There was a trend toward benefit in PFS and OS curves between the two groups. Although this study is an exploratory study, data from applied studies in the post-transplantation maintenance phase suggest that this immunotherapy may be termed as a new, better and safer option.

Therefore, the investigators conducted a multicenter, randomized, controlled study based on retrospective research to further explore and validate the safety and efficacy of Blinatumomab as a maintenance therapy after high-risk B-ALL allogeneic transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-65 years
2. Diagnosis with acute B-lymphoblastic leukemia (B-ALL) expressed CD19
3. High-risk group B-ALL
4. Have suitable hematopoietic stem cell donors
5. No dysfunction of vital organs

Exclusion Criteria:

1. CR/MRD negative before blinatumomab maintenance
2. Active hepatitis B
3. HIV-infected
4. Active infections; acute and chronic GVHD requiring systemic immunosuppressive therapy;
5. severe impairment of vital organ function
6. Those judged by the investigator to be unsuitable for participation in this trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
2-year Event-free survival | through study completion, an average of 2 year

SECONDARY OUTCOMES:
2-year relapse rate | through study completion, an average of 2 year